CLINICAL TRIAL: NCT07328646
Title: EFFECTIVENESS OF A BEHAVIOR CHANGE INTERVENTION AIMED AT INCREASING PHYSICAL ACTIVITY IN PATIENTS WITH PERIPHERAL ARTERY DISEASE UNDERGOING ENDOVASCULAR REVASCULARIZATION
Brief Title: BEHAVIOR CHANGE INTERVENTION AFTER ENDOVASCULAR REVASCULARIZATION IN PAD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Ayşe Adıgüzel Bayar, Physiotherapist, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Phd Thesis
Record Dates: First submitted 2025-12-27; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: BEHAVIOR CHANGE-BASED PHYSICAL ACTIVITY INTERVENTION IN PAD PATIENTS AFTER ENDOVASCULAR REVASCULARIZATION
Keywords: Peripheral Artery Disease; Endovascular Revascularization; Physical Activity; Exercise Therapy; Behavior Change; Walking Capacity; Physical Function; Sedentary Behavior; Quality of Life
MeSH Terms: conditions — Peripheral Arterial Disease; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Behavior Change Intervention Group (Experimental): Participants in this arm will receive a structured behavior change-based physical activity intervention following endovascular revascularization.
  Interventions: Behavioral: Behavior Change-Based Physical Activity Program
- Supervised Exercise Group (Active Comparator): Participants in this arm will receive a supervised exercise program following endovascular revascularization, without a structured behavior change component.
  Interventions: Other: Combined Behavior Change and Exercise Program
- Combined Intervention Group (Experimental): Participants in this arm will receive a combined intervention including both a behavior change-based.
  Interventions: Other: Supervised Exercise Program

INTERVENTIONS:
Behavioral: Behavior Change-Based Physical Activity Program — The program will include behavior change techniques such as goal setting, self-monitoring, action planning, motivational support, and education to promote physical activity and reduce sedentary time.
  Arms: Behavior Change Intervention Group
Other: Supervised Exercise Program — The supervised exercise program will consist of structured exercise sessions aimed at improving walking capacity and physical function.
  Arms: Combined Intervention Group
Other: Combined Behavior Change and Exercise Program — This intervention integrates behavior change techniques with supervised exercise to enhance physical activity adherence, walking capacity, physical function, and quality of life.
  Arms: Supervised Exercise Group

SUMMARY:
The study titled "Investigation of the Effect of a Behavior Change-Based Physical Activity Program in Patients with Peripheral Artery Disease Who Have Undergone Endovascular Revascularization" will be conducted by Specialist Physiotherapist Ayşe ADIGÜZEL BAYAR. The study is designed to investigate the effects of a structured physical activity program planned using behavior change techniques after endovascular revascularization on walking capacity, physical function, physical activity level and quality of life in patients with peripheral artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants

Aged between 50 and 80 years

Able to read, understand, and write Turkish

Scheduled to undergo endovascular revascularization for peripheral artery disease

Exclusion Criteria:

* Positive exercise stress test result

Presence of cognitive or intellectual impairment

Presence of musculoskeletal or neurological conditions that may interfere with physical activity performance or outcome assessment

Presence of unstable chronic disease

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-10-29 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported physical activity level (IPAQ total score) | Baseline, 6 weeks, 12 weeks
  Self-reported physical activity level will be assessed using the International Physical Activity Questionnaire (IPAQ). The primary outcome is the change in total physical activity level, expressed as MET-minutes per week, from baseline.

SECONDARY OUTCOMES:
Change in walking capacity (6-Minute Walk Test distance) | Baseline, 6 weeks, 12 weeks
  Walking capacity will be assessed using the 6-Minute Walk Test. The primary endpoint is the change in 6MWT distance (meters) from baseline.
Change in physical function (SPPB total score) | Baseline, 6 weeks, 12 weeks
  Physical function will be evaluated using the Short Physical Performance Battery (SPPB). The outcome is the change in SPPB total score from baseline.
Change in walking impairment (WIQ total score) | Baseline, 6 weeks, 12 weeks
  Walking impairment will be evaluated using the Walking Impairment Questionnaire (WIQ). The outcome is change in WIQ total score from baseline.
Change in quality of life (SF-12 PCS and MCS) | Baseline, 6 weeks, 12 weeks
  Quality of life will be assessed using the 12-Item Short Form Health Survey (SF-12). Outcomes include changes in Physical Component Summary (PCS) and Mental Component Summary (MCS) scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Aydın Özel Medinova Hastanesi, Efeler, Aydın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will not be shared due to ethical and privacy considerations, as well as the absence of explicit participant consent for data sharing. The study involves a relatively small sample size, which may increase the risk of participant re-identification. Data will be reported only in aggregate form in scientific publications.

REFERENCES:
- [Background] Gardner AW, Montgomery PS, Wang M, Shen B. Minimal clinically important differences in daily physical activity outcomes following supervised and home-based exercise in peripheral artery disease. Vasc Med. 2022 Apr;27(2):142-149. doi: 10.1177/1358863X211072913. Epub 2022 Feb 15. PMID 35164605